CLINICAL TRIAL: NCT01983033
Title: Drop it. The Impact of a Training Protocol Focused on Coping With Negative Repetitive Thinking on Cognitive and Behavioural Functioning of People Suffering From GAD or Minor or Moderate Depressive Disorder or Depressive Disorder in Remission
Brief Title: Training Protocol 'Drop it'. The Impact of a Training Protocol Focused on Coping With Negative Repetitive Thinking on Cognitive and Behavioural Functioning of People Suffering From GAD or Minor or Moderate Depressive Disorder or Depressive Disorder in Remission
Acronym: Drop It
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/708; B670201318392 (Other: Belgian registration number)
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Repetitive Negative Thinking; General Anxiety Disorder; Depressive Disorder; Depression; Anxiety Disorders; Worrying; Rumination
MeSH Terms: conditions — Generalized Anxiety Disorder; Depressive Disorder; Depression; Anxiety Disorders; Rumination Syndrome | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- active treatment condition (ATC) (Experimental): training protocol 'drop it'
  Interventions: Behavioral: Drop It training session
- waiting list control (Other): no treatment other than treatment as usual
  Interventions: Behavioral: treatment as usual

INTERVENTIONS:
Behavioral: Drop It training session — 8 training sessions in group, sessions of 90 minutes, 7 sessions weekly, plus 1 session after 1 month
  Arms: active treatment condition (ATC)
Behavioral: treatment as usual — 12 weeks of no intervention other than treatment as usual
  Arms: waiting list control

SUMMARY:
Repetitive negative thinking (RNT) plays an important role in different psychiatric disorders, such as depressive and anxiety disorders, complicated grief, posttraumatic stress disorders, anorexia nervosa. RNT is seen as a vulnerability factor in the onset, duration, severity and relapse of those disorders. Although there is a lot of theoretical research, it is unknown if a group training protocol addressing RNT has an additional effect on Treatment as Usual (TAU) of patients with GAD or Depressive disorder. Our hypothesis is that a training intervention will show a significant effect on declined RNT activity (measured by PSWQ and LARRS), reduced identification with worrying/rumination (measured by CFQ-13 and a Visual Analogue Scale), and reduced scores on metacognitions questionnaire (MCV Dutch version of the MCQ), when compared to TAU (medication, psychotherapy or a combination of both treatments). Further we expect that this effect on RNT will not be temporary and the beneficial effects will remain present over a longer time (9 months). Our third hypothesis claims that reduced RNT will have an effect on Quality of Life, self-esteem and depressive and anxiety scores (measured respectively by WHO-QoL, Rosenberg Self Esteem Questionnaire, BDI-II and STAI; all of them in Dutch version). Fourth hypothesis concerns the effect of the training in the functioning on a neurobiological level. Here we expect that the beneficial effects of training on RNT will increase top-down prefrontal (dorsolateral) cortical control over an overactive bottom-up limbic system. To examine these neurobiological effects, we apply a multimodal approach where we combine resting state fMRI, structural MRI such as diffuse tensor imaging (DTI), anterior spin labelling (ASL). Further, in our department we developed an audio critique task where participants hear different kinds of critique amongst some of negative valence which will be especially problematic for ruminative patients reflecting difficulties and differences these top-down/bottom-up processes when compared to a healthy control group at baseline. Further, we hypothesize that only when coping with RNT is successful these neuronal processes will normalize. We do not expect changes in the waiting list group.

To examine these clinical and neuronal effects, people suffering from GAD and/or depression will be allocated by randomisation to an active treatment condition (ATC) and a waiting list control group (WLC). All the participants will be patients treated by general practitioner, psychologist or psychiatrist. Training exists of 8 sessions in group (max 12 participants) on a weekly basis, except for the last session, which takes place after one month). During the training people will get information on RNT, they will be trained in re-allocation of their attention, will receive some basic ideas about becoming aware of dysfunctional thinking and learn coping strategies such as stimulus control and engaging in positive activity.

Assessments will take place before and after treatment for the ATC. The WLC will be measured at the start of the WLC and 12 weeks later. Measurement takes place by means of questionnaires and fMRI. During the fMRI, people will undergo a resting state paradigm and some tasks triggering RNT. 3 and 9 months after the group treatment, participants will be evaluated again on RNT by means of questionnaires. Participants in WLC will receive group treatment from the moment the parallel active treatment condition is ended (e.g. after 12 weeks). This group will be evaluated immediately after training and at 3 and 9 months follow-up.

At the end of the training, after the 8th session, two participants per run will be asked to cooperate in a qualitative in-depth interview. We are interested in linking results with the group training with some factors such as quantity of sessions, degree of active participation in between sessions. We are also interested in defining which interventions are perceived as most useful and if there is a link between disorder and the usefulness of some interventions.

ELIGIBILITY:
Inclusion Criteria:

* GAD
* depression or depression in remission

Exclusion Criteria:

* other psychiatric pathology than GAD or depression screened by senior psychiatrist by means of MINI and psychiatric anamnesis
* Abuse of alcohol, drugs or medication other than prescribed by GP or psychiatrist
* no consent to participate in measurement (questionnaire or fMRI- for fMRI: except medical contra-indications)
* Insufficient knowledge of the current language (Dutch)
* Acute or chronic suicidality
* Acute psychosis or manic depressive disorder
* Not able to commit for the 8 sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
change in repetitive negative thinking | at baseline, at the end of active treatment (12 weeks), at 3 months follow-up and at 9 months follow-up
  degree of repetitive negative thinking (PSWQ Dutch version)
change in repetitive negative thinking | at baseline, at the end of active treatment (12 weeks), at 3 months follow-up and at 9 months follow-up
  degree of repetitive negative thinking (LARRS)
change in repetitive negative thinking | at baseline, at the end of active treatment (12 weeks), at 3 months follow-up and at 9 months follow-up
  changes in metacognitions on RNT (MCV Dutch version of MCQ)
change in repetitive negative thinking | at baseline, at the end of active treatment (12 weeks), at 3 months follow-up and at 9 months follow-up
  degree of identification/disengagement (CFQ-13)
change in repetitive negative thinking | at baseline, at the end of active treatment (12 weeks), at 3 months follow-up and at 9 months follow-up
  degree of identification/disengagement (VAS)

SECONDARY OUTCOMES:
change in resting state fMRI | at baseline and at the end of active treatment (12 weeks)
  Structural MRI and DTI fMRI combined with critique paradigm
change in Quality of Life | two weeks before active treatment,12 weeks after the start of the active treatment, 3 months after follow-up and 9 months after follow-up
  WHO Quality of Life Dutch version
change in self-esteem | two weeks before active treatment,12 weeks after the start of the active treatment, 3 months after follow-up and 9 months after follow-up
  measured by Rosenberg Self Esteem Questionnaire Dutch version
change in depression and anxiety | two weeks before active treatment/waiting list, 12 weeks after active treatment/waiting list, follow-up 3 and 9 months after active treatment
  BDI-II, STAI Dutch versions
change in personality features | two weeks before active treatment/waiting list, 12 weeks after the start of the active treatment/waiting list
  using the TCI (Temperament and Character Inventory)

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium